CLINICAL TRIAL: NCT05302206
Title: Colonic Glucose vs. Saline Infusion on Hormone Secretion and Glycemic Excursions
Brief Title: Colonic Glucose vs. Saline Infusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Sanyuan Hu, Professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-228
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Gastrointestinal Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with ileostomy without type 2 diabetes (Experimental): colonic glucose or saline infusion via ileostomy
  Interventions: Dietary Supplement: colonic infusion
- patients with ileostomy with type 2 diabetes (Experimental): colonic glucose or saline infusion via ileostomy
  Interventions: Dietary Supplement: colonic infusion

INTERVENTIONS:
Dietary Supplement: colonic infusion — colonic glucose or colonic saline infusion

SUMMARY:
The distal ileum and proximal colon, where the glucagon-like peptide 1 (GLP-1) releasing cells predominate, are important organs in mediating glycemic control. The proximal colon is not easy to access and the correspond in vivo research remains to be difficult. The investigators intend to recruit subjects who underwent rectal surgery with simultaneous protective ileostomy and evaluate hormone secretion and glycemic excursions via ileostomy glucose or saline infusion, and quantify the glucose absorption rate within the proximal colon.

ELIGIBILITY:
Inclusion Criteria:

* Male and postmenopausal females aged 18 - 75 years
* Body mass index (BMI) 20 - 35 kg/m2
* With protective ileostomy due to benign or malignant rectal surgery

Exclusion Criteria:

* History of postoperative adjuvant chemotherapy
* Other significant illness, including epilepsy, cardiovascular or respiratory disease
* Impaired renal or liver function (as assessed by calculated creatinine clearance < 90 mL/min or abnormal liver function tests (> 2 times upper limit of normal range))
* Donation of blood within the previous 3 months
* Participation in any other research studies within the previous 3 months
* Females who are pre-menopausal
* Inability to give informed consent
* Vegetarians

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
serum or plasma GLP-1 changes during colonic infusion | 180 minutes
  concentration of serum or plasma GLP-1 (pmol/L)
serum or plasma GIP changes during colonic infusion | 180 minutes
  concentration of serum or plasma GIP (pmol/L)
serum or plasma ghrelin changes during colonic infusion | 180 minutes
  concentration of serum or plasma ghrelin (pg/ml)
serum or plasma c-peptide changes during colonic infusion | 180 minutes
  concentration of serum or plasma c-peptide (pmol/L)
serum or plasma insulin changes during colonic infusion | 180 minutes
  concentration of serum or plasma insulin (pmol/L)
serum or plasma glucagon changes during colonic infusion | 180 minutes
  concentration of serum or plasma glucagon (pmol/L)
glucose absorption capacity | 180 minutes
  estimated glucose absorption rate during colonic glucose infusion

CONTACTS AND LOCATIONS:
Overall Officials: Kexin Wang, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided